CLINICAL TRIAL: NCT02478775
Title: Dysregulation of Follicle Stimulating Hormone (FSH) in Obesity: Functional and Statistical Analysis
Brief Title: Dysregulation of FSH in Obesity: Functional and Statistical Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0474; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-06-23 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Fertility
Keywords: obesity; fertility; infertility; reproductive hormones
MeSH Terms: conditions — Obesity; Infertility | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Frequent Blood Sampling, Degarelix (Experimental): Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Degarelix (GnRH antagonist) blockade over a 2-day period. This arm was terminated due to Adverse Events and the study was continued with the Cetrorelix product.
  Interventions: Drug: Degarelix (GnRH antagonist); Drug: recombinant FSH
- Frequent Blood Sampling, Cetrorelix (Experimental): Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Cetrorelix blockade over a 2-day period.
  Interventions: Drug: recombinant FSH; Drug: Cetrorelix

INTERVENTIONS:
Drug: Degarelix (GnRH antagonist) — Day-1: Blood samples will be obtained every 10 minutes for 10 hours. After 10 hours of blood samples have been collected, the GnRH antagonist degarelix will be given subcutaneously.
  Other Names: Firmagon
  Arms: Frequent Blood Sampling, Degarelix
Drug: recombinant FSH — Day-2: Blood samples will again be obtained every 10 minutes for 10 hours. Repeated boluses of exogenous recombinant FSH (rFSH) will be given by IV during this 10 hour visit.
  Other Names: rFHS
Drug: Cetrorelix — Day-1: Blood samples will be obtained every 10 minutes for 10 hours. After 10 hours of blood samples have been collected, the GnRH antagonist Cetrorelix will be given subcutaneously.
  Other Names: Cetrotide
  Arms: Frequent Blood Sampling, Cetrorelix

SUMMARY:
Excess maternal weight, especially obesity, influences almost every aspect of fertility, from conception to problems during pregnancy. The investigators will use novel statistical methods to clarify the hormonal changes behind reproductive health conditions. A better understanding of reproductive hormonal changes in obese women may offer a way to identify new treatments.

DETAILED DESCRIPTION:
Hypothesis. Insufficient FSH (Follicle-stimulating hormone) pulsatility, as seen in obesity, results in inadequate folliculogenesis and reduced ovarian steroid and protein production.

AIM: To test the hypothesis that insufficient FSH pulsatility, as seen in obesity, results in inadequate folliculogenesis and reduced ovarian steroid and protein production. The investigators will determine if exogenous FSH administered in a pulsatile fashion results in a significant increase of ovarian hormones in obese women. Serial inhibin B and E2 levels will be measured in obese and normal weight women undergoing frequent blood sampling studies before and after GnRH (Gonadotropin-releasing hormone) antagonist blockade.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 to 39 years old with regular menstrual cycles every 25-40 days
* Body mass of 18.5 kg/m2-24.9kg/m2 (normal weight controls) or greater than 30.0 kg/m2 (obese group)
* Prolactin and thyroid-stimulating hormone (TSH) within normal laboratory ranges at screening
* Baseline hemoglobin >11 gm/dl.

Exclusion Criteria:

* Diagnosis of polycystic ovary syndrome (PCOS), defined by the 2003 Rotterdam criteria as suggested by 2012 NIH Workshop
* History of chronic disease affecting hormone production, metabolism or clearance or use of thiazolidinediones or metformin (known to interact with reproductive hormones)
* Use of hormones affecting hypothalamic-pituitary-gonadal (HPO) axis (such as hormonal contraceptives) within 3 months of entry
* Strenuous exercise (>4 hours of intense physical activity per week)
* Pregnancy
* Breast-feeding
* Current attempts to conceive
* Significant recent weight loss or gain

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Polotsky, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Clinical and Translational Research Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luu TH, Kuhn K, Bradford AP, Wempe MF, Wittenburg L, Johnson RL, Carlson NE, Kumar TR, Polotsky AJ. Effects of pulsatile intravenous follicle-stimulating hormone treatment on ovarian function in women with obesity. Fertil Steril. 2023 Oct;120(4):890-898. doi: 10.1016/j.fertnstert.2023.05.170. Epub 2023 Jun 3. PMID 37276947

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants were excluded after signing the consent.
Groups:
- Experimental: Frequent Blood Sampling, Degarelix: Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Degarelix (GnRH antagonist) blockade over a 2-day period. This arm was terminated due to Adverse Events and the study was continued with the Cetrorelix product.
- Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight: Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Cetrorelix blockade over a 2-day period.
  Normal weight participants = 18.5 to 24.9 BMI
- Experimental: Frequent Blood Sampling, Cetrorelix: Obese: Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Cetrorelix blockade over a 2-day period.
  Obese participants = BMI of >30
Period: Overall Study
Arm/Group | Experimental: Frequent Blood Sampling, Degarelix | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese
Started | 6 | 27 | 27
Completed | 6 | 27 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Frequent Blood Sampling, Degarelix: Investigators will assess the change in inhibin B levels following repeated bolus dosing of recombinant FSH (rFHS) following Degarelix (GnRH antagonist) blockade over a 2-day period. This arm was terminated due to Adverse Events and the study was continued with the Cetrorelix product.
  BMI = 18.5 to 24.9 BMI
- Total: Total of all reporting groups
Arm/Group | Experimental: Frequent Blood Sampling, Degarelix | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese | Total
Number analyzed (Participants) | 6 | 27 | 27 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.9) | 27.2 (4.7) | 31.9 (4.1) | 29.6 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 27 | 27 | 60
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 6 | 24 | 24 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 6 | 7
  White | 5 | 24 | 20 | 49
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 27 | 27 | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 22.5 (2.5) | 22.4 (1.5) | 37.7 (6.2) | 30.1 (8.9)
Weight [Mean (Standard Deviation); unit: kg] | 59.8 (4.2) | 61.1 (5.4) | 102 (19.3) | 81.6 (24.9)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Peak Inhibin B
Description: This is defined as the maximum hormone value during Day 1 of the study subtracted from the maximum hormone value during Day 2.
Time Frame: Every 10 minutes over 2 10-hour frequent blood sampling sessions.
Population: The Degarelix arm is excluded because no data was collected from those participants. The Degarelix arm was terminated due to adverse events and was replaced with the Cetrorelix arm.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese
Number analyzed (Participants) | 27 | 27
picograms/mL | 100.8 (73.7) | 38.8 (37.9)

2. Secondary Outcome: Peak Inhibin B Per Subject
Description: Peak inhibin B will be measured every 10 minutes during day 1 and day 2 of the study. The highest inhibin B value will be defined as the peak.
Time Frame: Every 10 minutes over 10 hours on Day 1 and Day 2 of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese
Number analyzed (Participants) | 27 | 27
picograms/mL
  Day 1 maximum | 103.5 (43.8) | 87.5 (45.3)
  Day 2 maximum | 226.5 (105.3) | 126.3 (52.5)

3. Secondary Outcome: Peak E2 Per Subject
Description: E2 will be measured every 10 minutes on Day 1 and Day 2 of the study. The highest E2 value will be designated as the peak E2 value.
Time Frame: Every 10 minutes over 10 hours of Day 1 and Day 2 of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/L
Arm/Group | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese
Number analyzed (Participants) | 27 | 27
pg/L
  Day 1 | 65.1 (58.0) | 72.5 (37.7)
  Day 2 | 137.7 (61.8) | 99.1 (41.6)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Experimental: Frequent Blood Sampling, Degarelix | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight | Experimental: Frequent Blood Sampling, Cetrorelix: Obese
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 5/6 | 0/27 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Frequent Blood Sampling, Degarelix (N=6) | Experimental: Frequent Blood Sampling, Cetrorelix: Normal Weight (N=27) | Experimental: Frequent Blood Sampling, Cetrorelix: Obese (N=27)
Delay of menses (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The Degarelix arm is excluded from outcome measure data because no usable data could be collected from those normal weight participants. There were no participants in this arm that were of high BMI. The Degarelix arm was terminated due to adverse events and was replaced with the Cetrorelix arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT02478775/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02478775/ICF_001.pdf